CLINICAL TRIAL: NCT01785381
Title: Randomized Controlled Trial: Added Value of Coordinator for the Management of Hip Fracture Patients in a Network of Public Hospitals in Brussels.
Brief Title: RCT: Added Value of Coordinator for the Management of Hip Fracture Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Nyaruhirira Innocent, MD, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRIS recherche 2012820690007
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, hip fracture, fractures, Bone density
MeSH Terms: conditions — Osteoporosis; Hip Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention): usual care
- Added value of coordinator (Other): Added value of coordinator
  Interventions: Other: Added value of coordinator

INTERVENTIONS:
Other: Added value of coordinator — Added value of coordinator
  Arms: Added value of coordinator

SUMMARY:
Introduction: Hip fracture due to osteoporosis is associated with an extremely high mortality morbidity and loss of quality of life. The risk of future fracture after a first hip fracture is increased. Several studies reported that patients who suffered from a fracture are not optimally treated and do not receive osteoporosis treatment after the first fracture episode.

Aim: To evaluate whether a coordinator increases the optimal management of osteoporotic fracture patients and hip fracture patients.

DETAILED DESCRIPTION:
Material and methods: Population: Identification in the "IRIS public hospital network of all patients above 50 years" who suffer from hip fracture. Exclusion of those due to high energy fractures and due to known cancer.

First observational phase of treatment followed by randomized controlled trials of 2 years.

Intervention (RCT): Added value of a coordinator. Measured outcomes : A. New fractures. B. A score of optimal management of osteoporosis.

Definition of the score and management: 1. Realization of a bone density measurement. 2. Identification of secondary osteoporosis. 3. Identification of risk factors and calculation of the probability of a future fracture using FRAX score. 4. Attempt to correct risk factors of osteoporosis when possible. 5. Prevention of falls. 6. Prescription of calcium and vitamin D. 7. Prescription of a medical osteoporosis treatment. 8. Report to the general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Identification in the "IRIS public hospital network of all patients above 50 years" who suffer from hip fracture.

Exclusion Criteria:

* Exclusion of those due to high energy fractures and due to known cancer.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
A score of optimal management of osteoporosis. | 3-6 months
  Definition of the score and management: 1. Realization of a bone density measurement. 2. Identification of secondary osteoporosis. 3. Identification of risk factors and calculation of the probability of a future fracture using FRAX score. 4. Attempt to correct risk factors of osteoporosis when possible. 5. Prevention of falls. 6. Prescription of calcium and vitamin D. 7. Prescription of a medical osteoporosis treatment. 8. Report to the general practitioner.

SECONDARY OUTCOMES:
New fractures. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRIS Hospitals, Brussels, Belgium